CLINICAL TRIAL: NCT03420846
Title: Efficiency of Presurgical Basal Cell Carcinoma Margin Mapping Using Optical Coherence Tomography
Brief Title: Efficiency of Presurgical Basal Cell Carcinoma Margin Mapping
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding exhausted. Sufficient data already collected.
Sponsor: Michelson Diagnostics Ltd. (Industry)
Collaborators: Skin Care Network Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1202
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to two arms. Participants in the first arm receive Mohs surgery using OCT mapping to delineate tumor margins.
  Participants in the Control Arm receive Mohs surgery using clinical estimation of tumor margins (ie. standard care) The average number of Mohs surgery cycles will be compared for the two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCT Mapped arm (Experimental): OCT is used to map the tumour margins as the first stage MMS estimate
  Interventions: Other: OCT Mapped
- Control arm (No Intervention): Standard MMS is performed

INTERVENTIONS:
Other: OCT Mapped — Presurgical mapping of Basal Cell Carcinoma margins
  Arms: OCT Mapped arm

SUMMARY:
This Interventional Randomised Controlled study is intended to establish that presurgical margin mapping of BCCs with OCT results in a reduction of the number of MMS surgery stages without adversely impacting clinical outcome, resulting in shorter patient stays and more efficient use of surgical and operating room resources.

DETAILED DESCRIPTION:
Basal Cell Carcinoma (BCC) is the most common malignancy in humans. Its incidence is continuously increasing. The head and neck areas are most commonly affected due to their increased lifetime exposure to sun compared to other body parts. BCC is often treated by surgical excision which has high cure rate compared to other treatment modalities, but leaves a visible scar which can affect the quality of life of the patient, depending on the location and size of the excision. Mohs Micrographic Surgery (MMS) was developed to minimize the size of the surgical excision whilst maintaining very high cure rate. The main drawback of MMS is that repeated surgery procedures are usually required to eliminate all of the tumour using specialist resources located at the clinic.

Optical Coherence Tomography (OCT) allows non-invasive in-vivo imaging of superficial skin lesions. It is in routine clinical use for diagnosis of BCCs, and the diagnostic sensitivity and specificity is well established in published multi-centre trials. A further potential application of OCT is the pre-surgical mapping of the lateral margins of BCC. If the margins of a BCC were accurately known prior to commencing an MMS treatment, the treatment could be performed much more quickly, resulting in shorter patient stays and more efficient use of surgical and operating room resources. Previously published research has already shown that OCT mapping of BCC margins is more accurate than clinical assessment; the objective of the present study is to demonstrate that pre-surgical mapping of BCC margins with OCT is also more efficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven BCCs who have been referred for MMS

Exclusion Criteria:

* Patients with BCCs larger than 6 cm2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Average number of Mohs stages | 1 day
  Is the average number of Mohs stages < 1.4 with a 95% confidence level. (P < 0.025)

SECONDARY OUTCOMES:
Size of the surgical defect | 1 day
  Validate that the reduction in MMS stages by use of OCT mapping does not result in an increase in the size of the surgical defect
Average time taken to perform OCT margin mapping | 1 day
  Show that the average time taken to perform OCT margin mapping is < 5 minutes for lesions of area < 2 cm2

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stevens, Principal Investigator — Skin Care Network Ltd.
Locations (1):
- SkinCare Network, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03420846/ICF_000.pdf
  • Study Protocol (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT03420846/Prot_001.pdf